CLINICAL TRIAL: NCT06748508
Title: A Multicenter, Prospective, Open-label, Randomized Controlled, Phase II Clinical Trial Comparing the Efficacy of Sintilimab Plus Nab-POF Regimen, Sintilimab Plus XELOX Chemotherapy, and Lenvatinib, Sintilimab Plus XELOX Chemotherapy in the Treatment of HER2-negative, Metastatic Gastric Cancer
Brief Title: Comparing the Efficacy of Sintilimab Plus Nab-POF Regimen, Sintilimab Plus XELOX Chemotherapy, and Lenvatinib, Sintilimab Plus XELOX Chemotherapy in the Treatment of HER2-negative, Metastatic Gastric Cancer
Acronym: FDZL-GC003
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Weijian Guo, chief physician, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MGC-NabPOF
Record Dates: First submitted 2024-12-03; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Gastric (Stomach) Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — sintilimab; lenvatinib; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- XELOX regimen plus sintilimab (Active Comparator): sintilimab 200mg ivgtt d1+oxaliplatin 130mg/m2 ivgtt d1+xeloda 1000mg/m2 bid po d1-14，q3w
  Interventions: Drug: Sintilimab, oxalipaltin, 5FU,Nab-paclitaxel,lenvatinib
- Nab-POF regimen plus sintilimab (Experimental): sintilimab (200mg for the first time, 100mg for the second time, in alteration) ivgtt d1+oxaliplatin 85mg/m2 ivgtt d1+Nab-paclitaxel 125 mg/m2 ivgtt d1+5FU 2.4g/m2 civ48h, q2w
  Interventions: Drug: Sintilimab, oxalipaltin, 5FU,Nab-paclitaxel,lenvatinib
- XELOX regimen plus sintilimab plus lenvatinib (Experimental): sintilimab 200mg ivgtt d1+oxaliplatin 130mg/m2 ivgtt d1+xeloda 1000mg/m2 bid po d1-14+lenvatinib 8mg(<60kg) or 12mg(≥60kg) po qd，q3w
  Interventions: Drug: Sintilimab, oxalipaltin, 5FU,Nab-paclitaxel,lenvatinib

INTERVENTIONS:
Drug: Sintilimab, oxalipaltin, 5FU,Nab-paclitaxel,lenvatinib — Patients were randomized in a 1:1:1 ratio to three treatment groups: control group A: pembrolizumab combined with XELOX regimen, the regimen was repeated every 3 weeks, and tumor efficacy was evaluated every 2 treatment cycles. Group B: treatment regimen was pembrolizumab combined with Nab-POF regimen, the regimen was repeated every 2 weeks, and tumor efficacy was evaluated every 3 treatment cycles. Group C: treatment regimen was pembrolizumab combined with XELOX regimen and lenvatinib, the regimen was repeated every 3 weeks, and tumor efficacy was evaluated every 2 treatment cycles.
  Other Names: xeloda

SUMMARY:
This trial is a prospective, open, randomized, phase II clinical study. It compares the current first-line treatment for advanced gastric cancer in phase II clinical trials, with the best efficacy being the combination of orient-16 study with sintilimab and XELOX regimen. The purpose of this study is to evaluate whether adding anti-angiogenic drugs or chemotherapy drugs on the basis of two-drug chemotherapy regimen (XELOX regimen) and PD-1 monoclonal antibody can improve efficacy for advanced gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged over than 18 years
2. Histologically or cytologically confirmed gastric adenocarcinoma (including GEJ adenocarcinoma)
3. Presence of measurable lesions(RECIST 1.1)
4. Newly diagnosed patients; or patients with recurrence after surgery, who have been off adjuvant chemotherapy for at least 6 months and have not received any anti-cancer treatment within the past 6 months
5. ECOG PS score: 0-1
6. Expected survival over than 3 months
7. Normal major organ function or reserve, meeting the following criteria (determined by laboratory test data within 7 days (inclusive) before screening): HB ≥90 g/dL, ANC ≥1.5×109/L, PLT ≥100×109/L; BIL<1.5×ULN, ALT and AST <2.5×ULN, if with metastases to liver, then ALT, AST <5×ULN; serum Cr≤1×ULN, endogenous creatinine clearance >50 mL/min (calculated by CK formula), international normalized ratio (INR) or prothrombin time (PT) ≤1.5×ULN, if the subject is receiving anticoagulant therapy, PT should be within the intended range of the anticoagulant drug
8. Subjects who voluntarily participate in this study, sign the informed consent form, have good compliance, and cooperate with follow-up

Exclusion Criteria:

1. Histopathological assessment of HER2 positivity (immunohistochemistry 3+ or immunohistochemistry 2+ and FISH positive)
2. Known dMMR/MSI-H
3. History of other malignant neoplasms within 3 years prior to enrollment, except for cured cervical carcinoma in situ or basal cell carcinoma
4. Presence of brain metastases to meninges
5. Malignant pleural or peritoneal effusion
6. Presence of gastrointestinal obstruction, gastrointestinal haemorrhage (fecaloccult blood +++ or higher), or perforation
7. Prior treatment with anti-PD-1, anti-PD-L1, or anti-PD-L2, CD137, CTLA-4 antibodies, or any other antibody or drug specifically targeting T-cell co-stimulatory or checkpoint pathways
8. Subjects with active or history of autoimmune diseases that might relapse (e.g., systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, autoimmune thyroid disorder, multiple sclerosis, vasculitis, glomerulonephritis, etc.), or high-risk patients (e.g., those requiring immunosuppression after organ transplant), except for those with vitiligo, psoriasis, alopecia, or Graves' disease that have not required systemic treatment within the past 2 years, or hypothyroidism requiring only thyroid hormone replacement therapy, or Type I diabetes mellitus requiring only insulin replacement therapy
9. Current interstitial lung disorder or pneumonia, pulmonary fibrosis, acute lung disorder, or radiation pneumonitis
10. Participation in other drug clinical studies within 4 weeks prior to the first dose (based on the use of investigational drug), except observational (non-interventional) clinical studies
11. Use of immunosuppressant drugs within 4 weeks prior to the first dose of study treatment, excluding nasal, inhaled, or other topical glucocorticoids or physiological doses of systemic glucocorticoids (i.e., no more than 10 mg/day of prednisone or equivalent dose of other glucocorticoids), or short-term (no more than 7 days) use of glucocorticoids for the prevention or treatment of non-autoimmune allergic diseases
12. Receipt of live attenuated vaccines within 4 weeks prior to the first dose of study treatment or planned immunization during the study period. Note: Inactivated seasonal influenza vaccines for injection are allowed within 4 weeks prior to the first dose; however, live attenuated influenza vaccines are not allowed.
13. Major surgery (craniotomy, thoracotomy, or laparotomy) within 4 weeks prior to the first dose of study treatment or anticipated need for major surgery (not related to this study) during the study treatment period.
14. History of human immunodeficiency virus (HIV) infection (i.e., HIV antibody positive), or other acquired or congenital immunodeficiency diseases, or history of organ transplant or stem cell transplant
15. Active chronic hepatitis B or active hepatitis C; hepatitis B virus carriers, but patients with stable hepatitis B viral loads after drug therapy (HBV DNA ≤ 200 IU/mL or copy number < 1000 copies/mL), and patients who have cleared hepatitis C virus (HCV RNA negative) are eligible for enrollment
16. Known active pulmonary tuberculosis
17. Patients with severe infection within 4 weeks before the first dose, or active infection requiring oral or vein antibiotic therapy within 2 weeks before the first dose
18. Symptomatic congestive cardiac failure (New York Heart Association Class II-IV) or symptomatic or poorly controlled arrhythmia
19. Uncontrolled hypertension (blood pressure systolic ≥160 mmHg or blood pressure diastolic ≥100 mmHg) despite standard treatment
20. Any arterial embolism event within 6 months before enrollment, including myocardial infarction, angina unstable, cerebrovascular accident, or transient ischemic attack
21. History of deep vein thrombosis, pulmonary embolism, or any other severe embolism within 3 months before enrollment (thrombosis originating from implanted venous access port or catheter, or superficial vein thrombosis is not considered as "severe" thromboembolism)
22. History of definite neurological or mental disorder: such as epilepsy, dementia, poor compliance, or peripheral nervous system disorders
23. Alcohol dependence or history of drug addiction or drug abuse within the past year
24. Pregnant or lactating women,women of childbearing potential who are not taking adequate contraception
25. Other acute or chronic disease, mental disorder, or laboratory test abnormality that might lead to the following results: increased risk associated with study participation or study drug administration, or interference with the interpretation of study results, and the investigator judges the patient to be ineligible for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Estimated)
Dates: Start 2024-12-25 (Estimated); Primary Completion 2027-07-25 (Estimated); Study Completion 2027-12-25 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | the duration from the date of randomization to any documented tumor progression or death due to any cause，assessed up to 24 months
  he proportion of patients whose tumor decrease to a certain size and remained for a certain period of time, including those with complete response (CR) and partial response (PR)

SECONDARY OUTCOMES:
Overall survival | the duration from the date of randomization to the date of death due to any cause,assessed up to 48 months
Progression-free survival time | the duration from the date of randomization to any documented tumor progression or death due to any cause, assessed up to 48 months
Disease control rate | the duration from the date of randomization to any documented tumor progression or death due to any cause, assessed up to 24 months
  assessed based on the RECIST 1.1 criteria, including complete response, partial response, and stable disease

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Fudan University Cancer Hospital, Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No